

Version Date: November 18, 2024

TO: ALL NATIONAL CLINICAL TRIALS NETWORK (NCTN) MEMBERS; CTSU

FROM: SWOG Network Operations Center (protocols@swoq.org)

RE: <u>\$1929</u>, "Phase II Randomized Study of Maintenance Atezolizumab Versus

Atezolizumab in Combination with Talazoparib in Patients with SLFN11 Positive

Extensive Stage Small Cell Lung Cancer (ES-SCLC)"

#### Revision #10

Study Chair: M.D.
Phone number: E-mail: S1929@swoq.org

#### **Action Codes**

- (√) Expedited review allowed
   (√) Patients Must be Informed\*
- (√) Consent Must Be Amended\*

\*See "Patient Notification and Use of Consent Addendum" and "Regulatory Considerations" instructions below.

# **Key Updates**

- (√) Informed Consent changes
- (√) Other: AE Reporting Table update
- ( √ ) Other: Talazoparib (NSC 771561) CAEPR updated

All sites: The protocol and/or informed consent form changes have been approved by the CIRB and must be activated within 30 days of distribution of this notice through the CTSU Bi-Monthly Broadcast email.

#### Revision # 10

S1929 has been revised with the following changes in response to a Request for Rapid Amendment (RRA) for Talazoparib (NSC 771561) from Dr. 2024. The associated Action Letter is attached. The AE table has been updated in response to CTEP's global safety update. The main change is the requirement for the 24-hour notification for ALL SAEs, irrespective of grade/severity, if the AEs meet any of the SAE criterion defined in FDA regulations, followed by a completed expedited report in 5 or 10 calendar days. The above referenced protocol has been revised as follows:

#### **Protocol Changes**

- The version date has been updated.
- The talazoparib drug ID has been updated to reflect the change in drug ownership, now Pfizer.
- Section 3.2c: This section has been updated with the most recent CAEPR for Talazoparib (PF-06944076) (Version 2.5 September 23, 2024). The following changes have been made to the Talazoparib CAEPR:
  - a. Increase in Risk Attribution:
    - i. Changed to Likely from Less Likely: Anorexia

4201 Medical Drive, Suite 250 | San Antonio, TX 78229 | OFFICE 210-614-8808 | FAX 210-614-0006





- ii. <u>Changed to Less Likely from Also Reported on Talazoparib Trials But With</u> Insufficient Evidence for Attribution: Dysgeusia
- b. Decrease in Risk Attribution:
  - i. Changed to Less Likely from Likely: Alopecia; Diarrhea; Headache; Vomiting
- 4. Section 8.7c, 8.7e, and 8.7g: These sections have been updated with the latest submission instructions and contact information.
- 5. Section 8.7e: This section has been updated with the most recent AE Reporting Table for late phase 2 and phase 3 studies (Effective date: August 30, 2024).

#### **Screening Consent Form Changes**

1. The version date has been updated. No additional changes have been made.

#### **Treatment Consent Form Changes**

- The version date has been updated.
- 2. The talazoparib drug ID has been updated to reflect the change in drug ownership, now Pfizer.
- 3. **Possible side effects of Talazoparib (PF-06944076):** The risk profile date has been updated to Table Version 2.5, September 23, 2024.
- 1. **"What risks can I expect..."** The following changes have been made to the Possible Side effects of Talazoparib (PF-06944076) risk section:
  - a. New Added Risk to Occasional:
    - i. Changes in taste
  - b. Increase in Risk Attribution:
    - i. Changed to Common from Occasional: Loss of appetite
  - c. <u>Decrease in Risk Attribution:</u>
    - i. Changed to Occasional from Common: Diarrhea, Vomiting, Headache, Hair loss

#### Patient Notification and use of Consent Addendum:

Please note that the information provided below regarding patient notification and amendments to local consent forms reflects SWOG's minimum requirements. Sites should refer to the policies/procedures of the IRB of record to determine whether they have any more stringent requirements.

SWOG has determined that the changes above that are **bolded** may affect a patient's willingness to participate in the study; therefore, SWOG requires that patients be notified of these changes.

#### Who must be informed?

All patients currently receiving on study treatment with Talazoparib (PF-06944076).

#### How must patients be notified?

• <u>For patients currently receiving Talazoparib (PF-06944076)</u>. Notification must take place either via the attached Consent Addendum or via amended consent form by next study visit. After the

change has been discussed with the patient, the patient must sign and date either the Consent Addendum or the 11/1/2024 version of the consent form.

What is the notification deadline and process?

- For patients currently receiving treatment with Talazoparib (PF-06944076): Patients must be notified by their next scheduled visit or within 90 days after CTSU distribution of this revision, whichever is sooner.
- CIRB has approved the attached Consent Addendum; therefore, the Consent Addendum may be utilized immediately to notify patients of these changes.

# Regulatory Considerations:

Do local consent forms need to be updated?

 It depends. If your site will utilize the updated consent form for notification and formal reconsent then local consent forms must be updated. If your site will not utilize updated consent form for notification and formal reconsent then local consent forms need not be updated.

The updated protocol and model informed consents, and consent addendum can be accessed from the CTSU website (<a href="www.ctsu.org">www.ctsu.org</a>). Please discard any previous versions of the documents and replace with the updated versions. Please contact mailto:lungquestion@crab.orgor 206/652-2267 with any questions.

This study has been reviewed and approved by the NCI's Central Institutional Review Board (CIRB).

This memorandum serves to notify the NCI, and SWOG Statistics and Data Management Center.

cc: PROTOCOL & INFORMATION OFFICE , M.D., M.S. , M.D., MPH

# <u>S1929</u> Research Study Informed Consent Document (Screening Consent)

**Study Title for Participants:** Testing Maintenance Therapy for Small Cell Lung Cancer in Patients with SLFN11 Positive Biomarker

# Official Study Title for Internet Search on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>:

<u>S1929</u>, "Phase II Randomized Study of Maintenance Atezolizumab versus Atezolizumab in Combination with Talazoparib in Patients with SLFN11 Positive Extensive Stage Small Cell Lung Cancer (ES-SCLC)" NCT#: 04334941

# Overview and Key Information (This section is a summary of the screening consent form)

#### What am I being asked to do?

We are asking you to take part in a research study. This study has public funding from the National Cancer Institute (NCI), part of the National Institutes of Health (NIH) in the United States Department of Health and Human Services. We do research studies to try to answer questions about how to prevent, diagnose, and treat diseases like cancer.

We are asking you to take part in this research study because you have extensive stage small cell lung cancer (ES-SCLC).

#### Taking part in this study is your choice.

You can choose to take part, or you can choose not to take part in this study. You also can change your mind at any time. Whatever choice you make, you will not lose access to your medical care or give up any legal rights or benefits.

This document has important information to help you make your choice. Take time to read it. Talk to your doctor, family, or friends about the risks and benefits of taking part in the study. It's important that you have as much information as you need and that all your questions are answered. See the "Where can I get more information?" section for resources for more clinical trials and general cancer information.



# Why is this study being done?

This study is being done to answer the following question:

Can we lower the chance of small cell lung cancer growing or spreading by adding talazoparib to the usual atezolizumab treatment?

We are doing this study because we want to find out if this approach is better or worse than the usual approach for small cell lung cancer. The usual approach is defined as care most people get for small cell lung cancer.

# What is the usual approach to treating small cell lung cancer?

The usual approach for patients who are not in a study is treatment with atezolizumab alone.

# What are my choices if I decide not to take part in this study?

- You may choose to have the usual approach described above.
- You may choose to take part in a different research study, if one is available.
- You may choose not to be treated for cancer.
- You may choose to only get comfort care to help relieve your symptoms and not get treated for your cancer.

#### What will happen if I decide to take part in the screening study?

If you decide to be screened for this study, we will ask you to submit a tumor sample which will be tested for the Schlafen family member 11 (SLFN11) protein at a special laboratory. The study doctor will discuss the screening test results with you. If the screening test shows the tumor sample is SLFN11 positive, you will be given another consent that explains the procedures and possible risks for the treatment study.

If the screening test shows the tumor sample is SLFN11 negative, you will not be able to go on to the treatment part of the study. Other treatment options will be discussed with you.

# What are the risks and benefits of taking part in the screening study?

There are both risks and benefits to taking part in the screening study. It is important for you to think carefully about these as you make your decision.



#### **Risks**

We want to make sure you know about a few key risks right now. We give you more information in the "What risks can I expect from taking part in the screening study?" section of this consent.

If you choose to take part in the screening study, there is a risk that the screening test used to detect SLFN11 protein may give the wrong results. These results may be a "false positive" or "false negative".

- False positive results will show that you do have the protein SLFN11, which, in fact, you do not have.
- **False negative** results occur when they show that you **do not** have the SLFN11 protein, which, in fact, you **do** have. This means that you would not be allowed to take part in the study, despite having the SLFN11 protein that should allow you to take part.

There may be some risks that the study doctors do not yet know about.

#### **Benefits**

Screening for SLFN11 may allow you to take part in the treatment study. Research has shown that having SLFN11 may increase the benefit of the study treatment. There is evidence that the study approach can stabilize cancer for longer than the usual approach alone. It is not possible to know now if the study drugs will extend your time without disease compared to the usual approach. The screening study will help the study doctors learn things that will help people in the future.

# If I decide to take part in the screening study, can I stop later?

Yes, you can decide to stop taking part in the study at any time.

If you decide to stop, let your study doctor know as soon as possible. It's important that you stop safely. If you stop, you can decide if you want to keep letting the study doctor know how you are doing.

Your study doctor will tell you about new information or changes in the study that may affect your health or your willingness to continue in the study.

#### Are there other reasons why I might stop being in the study?

Yes. The study doctor may take you off the study if:

- Your health changes and the study are no longer in your best interest.
- New information becomes available and the study is no longer in your best interest.
- You do not follow the study rules.
- For women: You become pregnant while on the study.
- The study is stopped by the National Cancer Institute (NCI), Institutional Review Board (IRB), Food and Drug Administration (FDA), or study sponsor (SWOG). The study sponsor is the organization who oversees the study.



S1929 Screening Consent Page 4 Version Date 11/18/2024

It is important that you understand the information in the informed consent before making your decision. Please read, or have someone read to you, the rest of this document. If there is anything you don't understand, be sure to ask your study doctor or nurse.

# What is the purpose of the screening study?

The purpose of the screening portion of this study is to identify if there is SLFN11 protein present in the cancerous tumor in your body. This is necessary to determine if you are eligible for the treatment study.

Another purpose of the screening study is for the study doctors to learn if checking for the SLFN11 protein is helpful in picking the right cancer treatments.

There will be about 323 people in the screening study.

# What are the study groups?

This study has a screening step. The purpose of this step is to test your tumor to find out if it has a protein, SLFN11. If it does and you meet all the study requirements, then you will be randomized to a study group for treatment.

If the screening test shows the tumor sample is SLFN11 negative, you will not be able to go on to the treatment part of the study. Other treatment options will be discussed with you.



Another way to find out what will happen to you during this study is to read the chart below. Start reading at the left side and read across to the right following the lines and arrows.



#### What exams, tests, and procedures are involved in the screening study?

Before you begin the study, your doctor will review the results of your exams, tests, and procedures. This helps your doctor decide if it is safe for you to take part in the study. If you join the study, you will have more exams, tests, and procedures to closely monitor your safety and health. Most of these are included in the usual care you would get even if you were not in a study.

Some exams, tests, and procedures are a necessary part of the research study but would not be included in usual care. Listed below are procedures that will be done for research purposes only.

# SLFN11 testing

Before you begin the study, a small piece of tumor sample, which was already removed by surgery or biopsy, will be sent to special laboratories for the study. Your tissue will be tested for the SLFN11 protein. This test is required for you to take part in the study. You and your study doctor will get the results of this testing. The results of this testing will determine if you will receive treatment on this study.

Your study doctor will need to use some of the tissue left over from your biopsy when you were diagnosed with cancer. The SLFN11 testing on this sample is a required part of the study



S1929 Screening Consent Page 6 Version Date 11/18/2024

because the presence of SLFN11 protein is needed to proceed to the main study. This sample will be tested for the presence of SLFN11, as described above.

# What risks can I expect from taking part in the screening study?

If you choose to take part in the screening study, there is a risk that the screening test used to detect SLFN11 protein may give the wrong results. These results may be a "false positive" or "false negative".

- False positive results will show that you do have the protein SLFN11, which, in fact, you do not have.
- **False negative** results occur when they show that you **do not** have the SLFN11 protein, which, in fact, you **do** have. This means that you would not be allowed to take part in the study, despite having the SLFN11 protein that should allow you to take part.

The screening study will use a sample of your tissue. Generally, your hospital will keep some of your tissue. This tissue may be used to help treat your cancer in the future. Because the screening study will need to use some of this tissue, there is a small risk that it could be used up.

You also may have the following discomforts:

- Spend more time in the hospital or doctor's office.
- Be asked sensitive or private questions about things you normally do not discuss.
- May not be able to take part in future studies.

# What are my responsibilities in the screening study?

If you choose to take part in this study, you will need to:

- Keep your study appointments.
- Tell your doctor about:
  - o all medications and supplements you are taking
  - o any side effects
  - o any doctors' visits or hospital stays outside of this study
  - o if you have been or are currently in another research study.

#### What are the costs of taking part in the screening study?

There is no cost to you or your insurance associated with this screening. However, if testing of the tumor sample shows that you are SLFN11 positive you will be offered participation in the treatment study.

You and/or your health plan/insurance company will need to pay for the costs of caring for your cancer while on treatment, including the cost of tests, procedures, or medicines to manage any side effects, unless you are told that certain tests are supplied at no charge. Before you decide to be in the study, you should check with your health plan or insurance company to find out exactly what they will pay for.



S1929 Screening Consent Page 7 Version Date 11/18/2024

Talk to your insurance provider and make sure that you understand what your insurance pays for and what it doesn't pay for if you take part in this clinical trial. Also, find out if you need approval from your plan before you can take part in the study.

Ask your doctor or nurse for help finding the right person to talk to if you are unsure which costs will be billed to you or your insurance provider.

You will not be paid for taking part in the screening study. The research may lead to new tests, drugs, or other products for sale. If it does, you will not get any payment.

# What happens if I am injured because I took part in the screening study?

If you are injured as a result of taking part in the screening study and need medical treatment, please talk with your study doctor right away about your treatment options. The study sponsors will not pay for medical treatment for injury. Your insurance company may not be willing to pay for a study-related injury. Ask them if they will pay. If you do not have insurance, then you would need to pay for these medical costs.

If you feel this injury was caused by medical error on the part of the study doctors or others involved in the study, you have the legal right to seek payment, even though you are in a study. Agreeing to take part in the screening study does not mean you give up these rights.

# Who will see my medical information?

Your privacy is very important to us. The study doctors will make every effort to protect it. The study doctors have a privacy permit to help protect your records if there is a court case. However, some of your medical information may be given out if required by law. If this should happen, the study doctors will do their best to make sure that any information that goes out to others will not identify who you are.

Some of your health information, such as your response to cancer treatment, results of study tests, and medicines you took, will be kept by the study sponsor in a central research database. However, your name and contact information will not be put in the database. If information from the screening study is published or presented at scientific meetings, your name and other personal information will not be used.



S1929 Screening Consent Page 8 Version Date 11/18/2024

There are organizations that may look at or receive copies of some of the information in your study records. Your health information in the research database also may be shared with these organizations. They must keep your information private, unless required by law to give it to another group.

Some of these organizations are:

- The study sponsor, SWOG, and any company supporting the study now or in the future. This would include any organization helping the company with the study.
- The NCI Central IRB, which is a group of people who review the research with the goal of protecting the people who take part in the study.
- The FDA and the groups it works with to review research.
- The NCI and the groups it works with to review research.
- The NCI's National Clinical Trials Network and the groups it works with to conduct research.

In addition to storing data in the study database, data from studies that are publicly funded may also be shared broadly for future research with protections for your privacy. The goal of this data sharing is to make more research possible that may improve people's health. Your study records may be stored and shared for future use in public databases. However, your name and other personal information will not be used.

Some types of future research may include looking at your information and information from other participants to see who had side effects across many studies or comparing new study data with older study data. However, right now we don't know what research may be done in the future using your information. This means that:

- You will not be asked if you agree to take part in the specific future research studies using your health information.
- You and your study doctor will not be told when or what type of research will be done.
- You will not get reports or other information about any research that is done using your information.

There are laws that protect your genetic information. However, there is a risk that someone could get access to your genetic information and identify you by name. In some cases, employers could use your genetic information to decide whether to hire or fire you. The study doctors believe the risk of this happening is very small. However, the risk may increase in the future as people find new ways of tracing information. For more information about the laws that protect you, ask your study doctor.



# Where can I get more information?

You may visit the NCI web site at <a href="http://cancer.gov/">http://cancer.gov/</a> for more information about studies or general information about cancer. You may also call the NCI Cancer Information Service to get the same information at: 1-800-4-CANCER (1-800-422-6237).

A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

| You can talk to the study doctor about any questions or concerns you he to report side effects or injuries. Contact the study doctor of study doctor[s]) at (insert telephone number). | (insert name |
|---|---|
| For questions about your rights while in this study, call the of organization or center) Institutional Review Board at number). | (insert name<br>(insert telephone |
| My signature agreeing to take part in the study | |
| I have read this consent form or had it read to me. I have discussed it my questions have been answered. I will be given a signed and dated agree to take part in the screening portion of the study. | |
| Participant's signature (or legally authorized representative) | |
| Date of signature | |
| Signature of person(s) conducting the informed consent discussion | on |
| Date of signature | |

